CLINICAL TRIAL: NCT03863470
Title: Study of Therapeutic Exercise in Acute Respiratory Failure to Improve Neuromuscular Disability Trial
Acronym: STAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Scott Halpern, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 831966
Record Dates: First submitted 2019-02-27; First posted 2019-03-05 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Critical Illness; Acute Respiratory Failure
Keywords: Early ICU mobility
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Intervention (Control) (No Intervention): There is no trial-driven approach to care. All hospitals contribute a minimum of 12 weeks of outcomes data prior to adopting the intervention. Pre-specified outcomes data will be electronically extracted for patients meeting eligibility criteria but there will be no attempt to influence delivery of usual care within the ICU. The length of the control phase will differ for each ICU cluster, depending on the sequence in which ICU-clusters are assigned to switch to the intervention phase.
- Early mobilization intervention (Active Comparator): The clinical team will set a standardized mobility goal for each patient during morning rounds and display the goal on the patient's door. A facilitator will be established in the ICU to communicate mobility goals and activities across clinical personnel shifts. Patient mobility scores will be displayed to clinical and administrative staff in the ICU via the ICU board.
  Interventions: Behavioral: Early mobilization intervention

INTERVENTIONS:
Behavioral: Early mobilization intervention — The intervention consists of 3 components: 1) A simplified mobilization goal (using the Surgical Optimal Mobility Score) will be defined during daily morning ward rounds and displayed on the doors of patients' rooms; 2) a facilitator will communicate to the care team regarding mobility goals; 3) clinicians will receive feedback on patient's mobility as mobility scores will be made available electronically on the ICU board - a dashboard for monitoring patient care in the ICU
  Arms: Early mobilization intervention

SUMMARY:
This is a stepped-wedge, cluster randomized, trial evaluating the effect of an early goal-directed mobilization intervention for ICU patients with acute respiratory failure within 12 medical and surgical ICUs across 4 hospitals in the University of Pennsylvania Health System. The investigators will conduct a 54-week trial to measure the effect of the intervention on multiple patient-centered outcomes of patient physical function and cognition, in addition to ICU and hospital length of stay and duration of mechanical ventilation compared to usual care.

DETAILED DESCRIPTION:
The STAND trial aims to measure the effect of an early goal-directed mobilization algorithm versus usual care for ICU patients with acute respiratory failure in the medical and surgical ICUs across University of Pennsylvania Health System (UPHS) with respect to patient-centered outcomes of patient physical function and cognition as well as multiple secondary clinical outcomes. To achieve this goal, the investigators will conduct a 54-week stepped-wedge, cluster randomized, trial to test the intervention during the course of providing usual care among a large and diverse population of patients admitted to 12 ICUs across 4 hospitals within UPHS. The intervention is an early mobilization protocol implemented during a patient's stay in the ICU. It involves three steps: 1) the clinical team will set a standardized mobility goal for each patient during morning rounds and display the goal on the patient's door; 2) a facilitator will be established in the ICU to communicate mobility goals and activities across clinical personnel shifts; 3) patient mobility scores will be displayed to clinical and administrative staff in the ICU via the ICU board. Approximately 1,500 adult patients with continuous mechanical ventilation for ≥48 hours (without interruption) and baseline independent ambulatory status will be enrolled. Participating ICUs will be randomized into 6 clusters of 2 ICUs each. Each ICU contributes a minimum of 12 weeks of data under the usual care control condition prior to implementing the early mobilization intervention. Then, using the stepped-wedge design, all ICUs will implement the intervention in 6-week intervals with the order and timing of implementation determined by random assignment. By the end of the trial, all ICUs will have utilized the intervention for at least 12 weeks. The primary outcome is peak patient activity level as measure by the ICU mobility score (IMS) at ICU discharge. Secondary outcomes include an array of clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old; AND
* Admission to 1 of 12 participating ICUs; AND
* Continuous mechanical ventilation for ≥ 48 hours (without interruption); AND
* Baseline independent ambulatory status

Exclusion Criteria:

* Admitting diagnosis of any of the following conditions:

  * Cardiopulmonary arrest
  * Raised intracranial pressure
  * Acute neurological admission diagnosis
  * Subarachnoid hemorrhage
  * Ischemic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1917 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Peak hour patient activity level | Within 48 hours of ICU discharge
  Peak hour patient activity level as measured by the ICU mobility score (IMS) at ICU discharge. IMS score ranges from 0 to 10.

SECONDARY OUTCOMES:
ICU mortality | From ICU admission to ICU discharge, approximately 3 days
  ICU Mortality
ICU length of stay | From ICU admission to ICU discharge, approximately 3 days
  ICU length of stay (days)
Hospital length of stay | From hospital admission to hospital discharge, approximately 5 days
  Hospital length of stay (days)
Duration of mechanical ventilation | From hospital admission to hospital discharge, approximately 5 days
  Duration of time spent on continuous mechanical ventilation (hours)
Duration of time spent in deep sedation | From hospital admission to hospital discharge, approximately 5 days
  Duration of time spent in deep sedation (hours)
Neurological function | From hospital admission to hospital discharge, approximately 5 days
  Composite measure of delirium and coma free days
Richmond Agitation-Sedation Scale (RASS) | From hospital admission to hospital discharge, approximately 5 days
  RASS score at time of first spontaneous breathing trial. RASS score ranges from -5 (unarousable) to +4 (combative); A score of 0 = alert and calm.

CONTACTS AND LOCATIONS:
Overall Officials: William Schweickert, MD, Principal Investigator — University of Pennsylvania School of Medicine - Pulmonary, Allergy, and Critical Care; Scott D Halpern, MD PhD, Principal Investigator — University of Pennsylvania School of Medicine - PAIR Center; Juliane Jablonski, DNP RN, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schweickert WD, Jablonski J, Bayes B, Chowdhury M, Whitman C, Tian J, Blette B, Tran T, Halpern SD. Structured Mobilization for Critically Ill Patients: A Pragmatic Cluster-randomized Trial. Am J Respir Crit Care Med. 2023 Jul 1;208(1):49-58. doi: 10.1164/rccm.202209-1763OC. PMID 36996413